CLINICAL TRIAL: NCT04493541
Title: A Phase 1b Randomized, Double-blind, Placebo-controlled Study to Assess the Safety and Pharmacokinetics of BMS-986256 in Participants With Active Cutaneous Lupus Erythematosus
Brief Title: A Study to Assess the Safety and Drug Levels of BMS-986256 in Participants With Active Cutaneous Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM026-027; 2019-004044-29 (EudraCT Number)
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Lupus Erythematosus, Cutaneous
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-986256 (Experimental)
  Interventions: Drug: BMS-986256
- Placebo (Placebo Comparator)
  Interventions: Other: BMS-986256 Placebo

INTERVENTIONS:
Drug: BMS-986256 — Specified Dose on Specified Days
  Arms: BMS-986256
Other: BMS-986256 Placebo — Specified Dose on Specified Days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and drug levels of BMS-986256 in participants with cutaneous lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

a) Must have one of following diagnoses: i) Meet European League Against Rheumatoid (EULAR)/American College of Rheumatology 2019 Classification Criteria for systemic lupus erythematosus (SLE) OR ii) Biopsy-proven acute cutaneous lupus erythematosus (ACLE), subacute cutaneous lupus erythematosus (SCLE), or discoid lupus erythematosus (DLE): Participants without a concurrent SLE diagnosis are eligible b) Active cutaneous lupus disease, defined as a modified Cutaneous Lupus Erythematosus Disease Area and Severity Index- Activity (mCLASI-A) score ≥ 6 c) Active cutaneous lupus skin lesion(s) amenable to biopsy

• Women of childbearing potential (WOCBP) and men must agree to follow instructions for method(s) of contraception, if applicable

Exclusion Criteria:

* Active severe or unstable neuropsychiatric SLE
* Active, severe Lupus Nephritis (LN)
* Any British Isles Lupus Assessment Group (BILAG) A or B, unless within the constitutional, musculoskeletal and/or mucocutaneous domains

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events (SAEs) | Up to 24 weeks
Incidence of Adverse Events (AEs) | Up to 20 weeks
Number of laboratory test abnormalities: Hematology | Up to 20 weeks
Number of laboratory test abnormalities: Urinalysis | Up to 20 weeks
Number of laboratory test abnormalities: Clinical Chemistry | Up to 20 weeks
Incidence of clinically significant changes in physical examination findings | Up to 20 weeks
Incidence of clinically significant changes in vital signs: Body temperature | Up to 20 weeks
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 20 weeks
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 20 weeks
Incidence of clinically significant changes in vital signs: Heart rate | Up to 20 weeks
Incidence of clinically significant changes in Electrocardiogram (ECG) parameters | Up to 20 weeks

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986256 | Up to 20 weeks
Time to maximum concentration (Tmax) of BMS-986256 | Up to 20 weeks
Trough observed plasma concentration (Ctrough) of BMS-986256 | Up to 20 weeks
Area under the concentration-time curve over the dosing interval (AUC (TAU)) of BMS-986256 | Up to 20 weeks
Maximum observed plasma concentration (Cmax) of metabolite BMT-271199 | Up to 20 weeks
Time to maximum concentration (Tmax) of metabolite BMT-271199 | Up to 20 weeks
Trough observed plasma concentration (Ctrough) of metabolite BMT-271199 | Up to 20 weeks
Area under the concentration-time curve over the dosing interval (AUC (TAU)) of metabolite BMT-271199 | Up to 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Berlin, Germany

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm